CLINICAL TRIAL: NCT02501499
Title: Breastfeeding Buddies: An Exploratory Evaluation Study of a Peer Support Program
Brief Title: Breastfeeding Buddies: An Exploratory Evaluation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Manulife Centre for Community Health Research (Other)
Collaborators: Wilfrid Laurier University (Other); Kitchener Downtown Community Health Centre (Unknown); Health Nexus Best Start (Unknown)
Responsible Party: Sponsor
Other Study IDs: Manulife
Record Dates: First submitted 2015-06-29; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breastfeeding Buddies participants: Mothers that participated in Me Breastfeed workshops. Half will have been in the education-only group and half will have a buddy/peer support person in addition to the workshop.
  Interventions: Other: Breastfeeding Buddies
- Volunteer Focus Group: Breastfeeding buddies volunteers that deliver education and support programs.

INTERVENTIONS:
Other: Breastfeeding Buddies — a 2 hour breastfeeding workshop and if mother chooses, she is matched with a buddy who will contact her and offer breastfeeding support
  Groups: Breastfeeding Buddies participants

SUMMARY:
This is an exploratory, qualitative evaluation study of the Breastfeeding Buddies (BFB) program. The Breastfeeding Buddies Program is a peer-based education and support program offered through the Kitchener Downtown Community Health Centre. The KDCHC has received funding to undertake a qualitative exploratory study of the BFB program. KDCHC has partnered with researchers at the Manulife Centre for Community Health Research at Wilfrid Laurier University to plan and implement this study.

The purpose of the evaluation study is to understand the perspectives and experiences of Breastfeeding Buddies (BFB) participants and volunteers. The evaluation will explore the process of implementation of the BFB education and support programs and assess the program impacts from the perspective of participants and volunteers. The methods in this study are qualitative because the BFB program has never collected qualitative data from program participants and volunteers. In the past, evaluation of the program has been limited to pre and post surveys. This qualitative study includes two components:

1. Interviews 6-8 weeks after the participants due dates with consenting mothers who participated in the Me Breastfeed workshop - 10-12 mothers who were matched with a Buddy (optional for all workshop participants) will be interviewed and 10-12 mothers who did not seek a match (but did participate in the workshop) will be interviewed to explore what they learned, what was helpful and how the program can be improved.
2. One focus group with 10-15 Breastfeeding Buddies volunteers to explore the experiences and perspectives of the BFB volunteers.

DETAILED DESCRIPTION:
Breastfeeding has been demonstrated to offer numerous physical and emotional health benefits to infant and mother and is the recommended approach to infant feeding by all levels of health authorities. Canadian statistics reveal 89% of mothers initiate breastfeeding at birth but only 51% continue to do so when an infant has reached four months of age. Research has indicated that engaging informed, supportive peers and supportive communities may be effective methods to help mothers who wish to continue to breastfeed overcome common challenges.

This study seeks to explore the benefits and challenges in a Canadian peer support program. The study will assist the BFB to improve their programs and contribute to the growing body of research exploring breastfeeding interventions.This is an exploratory, qualitative evaluation study of the Breastfeeding Buddies (BFB) program.

BFB Program Description:

The Breastfeeding Buddies Program was initiated by breastfeeding mothers in the community and has been supporting breastfeeding families in Waterloo Region since 2003. Recognizing the value of mother-to-mother breastfeeding support, the aim of the Breastfeeding Buddies Program is to help increase the number of moms achieving success in breastfeeding through feeling connected and supported in their community. An informed decision making model is used and diversity is valued when supporting families. This peer based breastfeeding support is a partnership between the Kitchener Downtown Community Health Centre and Region of Waterloo Public Health and is available to all women in Waterloo Region.

Breastfeeding Buddies are matched with breastfeeding moms who have had similar experiences or may speak the same language and provide ongoing telephone support and share community resources. BFB's also regularly attend established community sites (e.g. Breastfeeding cafes at Early Years Centres) to provide support to moms on a drop-in basis. Initial contacts between BFBs and mothers are established prenatally when possible through the program coordinator, but may occur at any time in their breastfeeding experience. The program also offers a free 2 hour prenatal breastfeeding class called "Me? Breastfeed?" that is taught by BFBs. This practical workshop offers women and their partner's information on the first 7 days after birth, help with overcoming common challenges and community resources.

All Breastfeeding Buddy volunteers have successfully breastfed for at least 6 months (though many have breastfed for over one year), and are passionate about breastfeeding. They receive 20 hours of expert training with a nurse/lactation consultant and participate in monthly meetings to learn new skills.

The purpose of the evaluation study is to understand the perspectives and experiences of Breastfeeding Buddies (BFB) participants and volunteers.

The evaluation will explore the process of implementation of the BFB education and support programs and assess the program impacts from the perspective of participants and volunteers. The methods in this study are qualitative because the BFB program has never collected qualitative data from program participants and volunteers. In the past, evaluation of the program has been limited to pre and post surveys. This qualitative study includes two components:

1. Interviews 6-8 weeks after the participants due dates with consenting mothers who participated in the Me Breastfeed workshop - 10-12 mothers who were matched with a Buddy (optional for all workshop participants) will be interviewed and 10-12 mothers who did not seek a match (but did participate in the workshop) will be interviewed to explore what they learned, what was helpful and how the program can be improved.
2. One focus group with 10-15 Breastfeeding Buddies volunteers to explore the experiences and perspectives of the BFB volunteers.

ELIGIBILITY:
Inclusion Criteria:

* participated in Breastfeeding Buddies programs
* live birth
* consented to contact
* biological mother

Exclusion Criteria:

* less than age 16

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women will be recruited through the Me Breastfeed workshops. It is a self-selected community program that serves the Region of Waterloo (about 500,000 people and 6000 births a year). Workshops are offered twice monthly and have about 20 participants at each session.
  Mothers will be invited to participate in an interview 5-8 weeks past their indicated due date.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Mothers Experiences Interview | 2-3 months after participation in workshop (approximately 6 weeks past indicated due date of birth)
  An interview guide has been developed to assess the mother's experience and perspectives related to the intervention (education and/or support program). Questions are measuring whether the program is meeting it's intended goals including increasing knowledge, support, links to resources and increased initiation and duration of breastfeeding. The questions related to breastfeeding are based on a measure recently developed by health units in Ontario, Canada that is being used to monitor breastfeeding rates across the Province (Infant Feeding Surveillance Pilot Study). The survey is semi-structured in that the interviewer will be trained to probe participants to expand on their answers or ask relevant follow-up questions.

SECONDARY OUTCOMES:
Volunteer Focus Group Guide | 2 months after first workshop within study period
  A series of questions have been devised to explore the experiences of peer support volunteers to understand their perspectives as peer support volunteers, collect stories of successes, challenges and areas for improvement in the program.

REFERENCES:
- [Background] Jolly K, Ingram L, Khan KS, Deeks JJ, Freemantle N, MacArthur C. Systematic review of peer support for breastfeeding continuation: metaregression analysis of the effect of setting, intensity, and timing. BMJ. 2012 Jan 25;344:d8287. doi: 10.1136/bmj.d8287. PMID 22277543
- See also: Breastfeeding Statistics in Canada — http://www.statcan.gc.ca/pub/82-624-x/2013001/article/11879-eng.htm